CLINICAL TRIAL: NCT06511518
Title: Making Cognitive Behavioral Therapy for Cancer-related Fatigue Fit for Implementation in Patients With Cancer Receiving Palliative Systemic Treatment
Brief Title: Cognitive Behavioral Therapy for Cancer-related Fatigue in Patients With Cancer Receiving Palliative Systemic Treatment
Acronym: TIRELESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Hans Knoop, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL85495.018.23
Record Dates: First submitted 2024-02-23; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cancer; Palliative Treatment
MeSH Terms: conditions — Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benchmark study (Other): The results will be compared with those of a benchmark study, i.e. historical cohort of the same target group who received face-to-face CBT provided by psychologists in the TIRED study.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioural therapy (CBT) is a therapy that can help you manage your problems by changing the way you think and behave.

SUMMARY:
Cancer-related fatigue is highly prevalent in patients with cancer receiving palliative treatment and is experienced as one of the most burdensome symptoms affecting patients' daily functioning and quality of life. From the KWF-sponsored TIRED trial, we concluded that cognitive behavioral therapy (CBT) is effective in reducing fatigue in cancer patients with severe fatigue during palliative systemic treatment. However, in its current form, integration in routine medical care is difficult and scalability is a problem, as the intervention is time-intensive, requires face-to-face consults with a psychologists, and the availability of trained psychologists is limited.

The goal of this interventional study is to integrate interdisciplinary web-based CBT (inter-CBT) into clinical practice and prove non-inferiority in achieving a reduction in fatigue compared to face-to-face- CBT in patients with cancer receiving palliative treatment.

The main aims to answer are:

* To determine the non-inferiority of inter-CBT, compared to a benchmark study where CBT was provided by psychologists in its effect on reduction in cancer-related fatigue.
* To adapt CBT delivery to the needs of patients treated with palliative intent (interdisciplinary web-based CBT for cancer-related fatigue.
* To investigate its feasibility by evaluating the practical workability, acceptability, and burden for patients and health care providers.

Participant will follow the 12 weeks CBT intervention online, mainly guided by their nurse. Participants will start with a face-to-face session with the psychologists, partly together with their nurse, to start with setting their treatment goals. Then, they will work on the modules that are applicable to them. During the CBT intervention there will be a face-to-face session with their nurse to discuss the progress of their goals. Finally, all participants will complete the therapy by realizing their treatment goals. The outcomes with respect to fatigue severity and participants' goals will be discussed by the nurse with the participant in the final, face-to-face sessions. The face-to-face sessions will take 30 to max. 45 minutes, except for the first session, which will take one hour of which the nurse will be present during 15 minutes.

Researchers will compare the outcomes of the study to a benchmark study where CBT was provided by psychologists in its effect on reduction in cancer-related fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Receive systemic treatment with palliative intent for a solid tumor.
* Treatments include chemotherapy, targeted therapy, immunotherapy, and hormone therapy, possibly combined with surgery and/or radiation therapy
* Are ≥18 years old
* Are proficient in Dutch
* Report severe fatigue (Checklist Individual Strength, fatigue severity subscale [CIS-fatigue] score ≥35) with no known somatic explanation other than cancer and/or cancer treatment
* A life expectancy of ≥6 months according to their oncologist
* Access to a device with internet.

Exclusion Criteria:

* Symptomatic brain metastases
* Have a poor performance status (Karnofsky <70)
* Are currently receiving treatment for a mental disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity will be measured using the subscale fatigue severity (8 items, 7-point Likert scale) of the Checklist Individual Strength (CIS-fatigue). | Screening, baseline (T0), week 14 after T0 (T1) and week 26 after T0 (T2)
  The CIS-fatigue has shown to be sensitive to change, has good reliability and discriminative validity. Scores range from 8 to 56. A score of ≥35 indicates severe fatigue. Change = (week 14 score - baseline score).

SECONDARY OUTCOMES:
Fatigue will be assessed with the symptom scale Fatigue ((3 items, 4-point Likert scale) of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30, version 3.0). | Baseline (T0), week 14 after T0 (T1) and week 26 after T0 (T2)
  The EORTC QLQ-C30 is developed for use in clinical trials in cancer patients. Total scores on each subscale are linearly converted to a 0 to 100 scale. Higher scores indicate more fatigue. Change = (week 14 score - baseline score).
Quality of Life will be measured using the subscale global health status/QoL (2 items, 7-point Likert Scale) of the EORTC QLQ-C30. | Baseline (T0), week 14 after T0 (T1) and week 26 after T0 (T2)
  The EORTC QLQ-C30 is one of the most commonly used HRQoL instruments in the palliative setting and is known to be a reliable and valid measure of the quality of life of patients with cancer. A high score indicates good HRQoL. Change = (week 14 score - baseline score).
Functional impairment will be measured using the subscales emotional functioning (4 items, 4-point Likert scale) and physical functioning (5 items, 4-point Likert scale, range 0 to 100) of the EORTC QLQ-C30. | Baseline (T0), week 14 after T0 (T1) and week 26 after T0 (T2)
  Raw scores for both subscales are convertible to a score of 0 to 100. A high score represents a high level of functioning. Change = (week 14 score - baseline score).
Functional impairment will be assessed with the work and social adjustment scale (WSAS) | Baseline (T0), week 14 after T0 (T1) and week 26 after T0 (T2)
  Raw scores for both subscales are convertible to a score of 0 to 100. A high score represents a high level of functioning. Change = (week 14 score - baseline score).
Healthcare consumption | Baseline (T0), week 14 after T0 (T1) and week 26 after T0 (T2)
  In order to estimate the healthcare costs related to fatigue we will compare the therapist time spent per patient within the TIRELESS project with the time spent per patient within the benchmark study (TIRED study).
  We will use an adapted version of a questionnaire on health consumption and productivity loss (TiC-P). At baseline, patients will be asked about their healthcare consumption over the past 4 months.The healthcare consumption during the four months of the intervention (study participation) will then be compared to the four months preceding the intervention. A group of 25 patients who are severely fatigued and eligible for study participation, but who do not want to participate will be asked if they are willing to complete the TiC-P at the same time points (T0, T1, T2) as the study participants. We then will compare health care consumption of these two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Psychology, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Poort H, Verhagen CA, Peters ME, Goedendorp MM, Donders AR, Hopman MT, Nijhuis-van der Sanden MW, Berends T, Bleijenberg G, Knoop H. Study protocol of the TIRED study: a randomised controlled trial comparing either graded exercise therapy for severe fatigue or cognitive behaviour therapy with usual care in patients with incurable cancer. BMC Cancer. 2017 Jan 28;17(1):81. doi: 10.1186/s12885-017-3076-0. PMID 28129746
- See also: TIRED trial, the benchmark study — https://bmccancer.biomedcentral.com/articles/10.1186/s12885-017-3076-0